CLINICAL TRIAL: NCT07246681
Title: Role of Lignin in Treatment of Helicobacter Pylori Infection: A Double-blind Placebo-controlled Study
Brief Title: Lignin in Treatment of Helicobacter Pylori Infection
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Collaborators: EVERGREEN MEDICAL COMPANY (Unknown); Kafrelsheikh University (Other); Al-Azhar University, Egypt (Unknown); Ain Shams University, Egypt (Unknown); Security Forces Hospital Riyadh, Saudi Arabia (Unknown); Alyousif Hospital, Alkhobar, Saudi Arabia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-784
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter Pylori; Lignin; Eradication; Side effects

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): This is the study group who will receive the standard triple (proton pump inhibitor, amoxicillin, clarithromycin) therapy plus the hydrolyzed lignin 400 mg
  Interventions: Drug: Hydrolyzed Lignin
- Group II (Placebo Comparator): This is the study group who will receive the standard triple therapy (proton pump inhibitor, amoxicillin, clarithromycin) plus the placebo identical in color, shape, and taste with the hydrolyzed lignin
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydrolyzed Lignin — The drug will be supplied randomly to the group I
  Arms: Group I
Other: Placebo — Will be supplied randomly to Group II
  Arms: Group II

SUMMARY:
The goal of this clinical trial is to learn if drug hydrolyzed lignin works to treat H pylori infection in adults. It will also learn about the safety of drug lignin n the sitting of H pylori infection, and if it halts the side effects associated with H pylori triple therapy. The main questions it aims to answer are:

* Does drug hydrolyzed lignin improve the H pylori eradiation rate when it is added to the standard triple therapy used in treatment of H pylori?
* What medical problems do participants experience when taking drug hydrolyzed lignin? Researchers will compare drug hydrolyzed lignin to a placebo (a look-alike substance that contains no drug) to see if drug hydrolyzed lignin works to treat H pylori.

Participants will:

* Take drug hydrolyzed lignin or a placebo every day for 2 weeks beside the standard triple therapy
* Visit the clinic once every 1 week for checkup and questionnaire filling
* Check for H pylori eradication after treatment

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults, older than 18.
* Gender: all
* Patient with confirmed diagnosis of H pylori for the first time
* H pylori treatment naive patients
* Welling to participate

Exclusion Criteria:

* Patients with failed H pylori eradication
* Allergy to the used medications
* Patients with other structural bowel diseases e.g. celiac disease, ischemic colitis, IBD, chronic diarrhea
* General debilitating diseases e.g. decompensated cirrhosis, renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 2 weeks of continuous treatment, followed by 2 weeks of treatment and then testing again for presence\absence of the infection
  How much the H pylori eradication rate following the treatment

SECONDARY OUTCOMES:
Safety profile | up to 4 weeks (2 weeks active treatment and 2 weeks after treatment)
  The side effects related to the used medications (triple therapy and lignin)

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1- Öztekin M, Yılmaz B, Ağagündüz D, Capasso R. Overview of Helicobacter pylori Infection: Clinical Features, Treatment, and Nutritional Aspects. Diseases. 2021 Sep 23;9(4):66. doi: 10.3390/diseases9040066. PMID: 34698140; PMCID: PMC8544542. 2- Malfertheiner P, Megraud F, Rokkas T, Gisbert JP, Liou JM, Schulz C, Gasbarrini A, Hunt RH, Leja M, O'Morain C, Rugge M, Suerbaum S, Tilg H, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study group. Management of Helicobacter pylori infection: the Maastricht VI/Florence consensus report. Gut. 2022 Aug 8:gutjnl-2022-327745. doi: 10.1136/gutjnl-2022-327745. Epub ahead of print. PMID: 35944925. 3- Maldonado-Carmona N, Marchand G, Villandier N, Ouk TS, Pereira MM, Calvete MJF, Calliste CA, Żak A, Piksa M, Pawlik KJ, Matczyszyn K, Leroy-Lhez S. Porphyrin-Loaded Lignin Nanoparticles Against Bacteria: A Photodynamic Antimicrobial Chemotherapy Application. Front Microbiol. 2020 Nov 17;11:606185. 4- Sugiarto S, Leow Y, Tan CL, Wang G, Kai D. How far is Lignin from being a biomedical material? Bioact Mater. 2021 Jun 26;8:71-94. doi: 10.1016/j.bioactmat.2021.06.023. 5- Syed Waqas Ali Shah, Qi Xu, Muhammad Wajid Ullah, Zahoor, Sivasamy Sethupathy, Gabriel Murillo Morales, Jianzhong Sun, Daochen Zhu, Lignin-based additive materials: A review of current status, challenges, and future perspectives, Additive Manufacturing, Volume 74, 2023, 103711, ISSN 2214-8604, https://doi.org/10.1016/j.addma.2023.103711.(https://www.sciencedirect.com/science/article/pi). 6- Hunt R., Xiao S., Megraud F., Leon-Barua R., Bazzoli F., Van Der Merwe S., et al. (2011) Helicobacter pylori in developing countries. World Gastroenterology Organisation Global Guideline. J Gastrointestin Liver Dis 20: 299-304. 7- Alsohaibani F, Peedikayil M, Alshahrani A, Somily A, Alsulaiman R, Azzam N, Almadi M. Practice guidelines for the management of Helicobacter pylori infection: The Saudi H. pylori Working Group recommendations. Saudi J Gastroenterol. 2023 Nov-